CLINICAL TRIAL: NCT03158766
Title: Subclinical Propionibacterium Acnes Infection Estimation in the Intervertebral Disc (SPInE-ID): a Prospective Cohort
Brief Title: Subclinical Propionibacterium Acnes Infection Estimation in the Intervertebral Disc (SPInE-ID)
Acronym: SPInE-ID
Status: Completed | Type: Observational
Sponsor: Hospital Israelita Albert Einstein (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2998-17
Record Dates: First submitted 2017-05-15; First posted 2017-05-18 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2020-02

CONDITIONS: Infection; Intervertebral Disc Herniation; Propionibacterium Infection; Spinal Diseases; Discitis
Keywords: infection; intervertebral disc; Propionibacterium acnes; spine
MeSH Terms: conditions — Infections; Intervertebral Disc Displacement; Spinal Diseases; Discitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Lumbar Intervertebral Disc, Flavum ligament, Multifidus muscle
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Microdiscectomy: Patients with lumbar disc herniation who failed conservative treatment undergoing surgical treatment through microdiscectomy.
  Interventions: Other: Microdiscectomy

INTERVENTIONS:
Other: Microdiscectomy — It will be an observational study without interventions. Subjects with diagnose of lumbar disc herniation undergoing open decompression surgery (microdiscectomy) will be included and analyzed. There will be no direct intervention to the patient proposed by the study.

SUMMARY:
Subclinical infection of the intervertebral disc after lumbar disc herniation surgery has been correlated to chronic low back pain and vertebral endplate changes. The most commonly reported agent is Propionibacterium acnes. However, the real incidence is unclear, as it has been reported in some series ranging from 3.7% to 46%. Recently, a systematic review concluded that there is a relationship between P. acnes and endplate changes, but, there are so far no studies to verify whether the reported presence of that pathogen in the intervertebral discs is due to local infection or whether intraoperative contamination occurred during the collection of samples.

Thus, the main objective of this study is to estimate the incidence of subclinical infection in patients surgically treated for lumbar disc herniation.

To this end, a prospective cohort study will be conducted with a minimum of 95 patients between 18 and 65 years of age who have been submitted to surgery after failure of conservative treatment. The extruded disc will be removed and cultured for bacterial identification. As controls, the ligamentum flavum and the multifidus muscle, taken respectively before and after removal of the herniated fragment will also be cultured. Patients will be followed-up for a year and MRI will be done at the end of this period.

DETAILED DESCRIPTION:
INTRODUCTION Low back pain is a frequent condition in the population, as well as vertebral endplates abnormalities, described by Modic et al.(1,2), that affect up to 6% of the general population, and, up to 46% of patients with low back pain(3). Modic type I changes are described as vertebral bone marrow edema related to acute low back pain(4). When Modic changes are detected, chances of one presenting unspecific low back pain are 4.5 times higher(1,2).

Subclinical infection caused by low-virulence pathogen can possibly lead to vertebral endplate abnormalities, detected in magnetic resonance imaging (MRI) studies, and differentiation between infection and Modic changes may be difficult(5,6). Subclinical infection can also be associated with increasing low back pain(7). Albert et al(8) reported 61 patients who had undergone surgical treatment for lumbar disc herniation where 46% of cases had a positive culture. The same authors also reported that 80% of patients with a positive culture for anaerobic pathogens presented Modic type I changes at the adjacent vertebra after a two-year follow-up, against 44% of patients with negative culture. Some studies demonstrated the presence of low-virulence pathogens in intervertebral disc tissue cultures(6-10), most commonly reported to Propionibacterium acnes.

Chronic low back pain and Modic type I changes have been treated with antibiotics for up to 100 days with superior outcomes compared to sham treatment(7). Patients were treated with amoxicillin/clavulanate (500mg/125mg)(7) based on the study where sciatica is associated with Propionibacterium acnes(8).

However, Carricajo et al(11) suggest that the presence of P. acnes in the intervertebral discs is due to either external surgical or laboratory contamination. These authors detected positive disc culture in only 3.7% of cases out of 54 patients. Furthermore, same authors demonstrated that samples of spinal muscle and ligamentum flavum collected intraoperatively at the end of procedure had positive cultures in 14.8% of cases with a negative disc culture.

A systematic review performed by Urquhart et al(12) concluded, that there is moderate evidence that a relationship between positive culture with Modic type I changes and low back pain exists, although there was low evidence for relationship of cause. For that, authors concluded that new studies should be made to determine whether pathogens in the disc are originated from external contamination or if they are truly involved in the development of chronic back pain.

HYPOTHESIS Lumbar disc herniation is related to subclinical infection of the intervertebral disc Null hypothesis: incidence of subclinical infection is the same as incidence of cases without infection in patients with lumbar disc herniation treated with surgery.

OBJECTIVES Main purpose of this study is to identify if the presence of a infection pathogen in the intervertebral disc is real or if it is intraoperative contamination.

Secondary objectives are to analyze clinical prognostic factors in patients and diagnosis of infection.The study also proposes to analyze the relationship between radiological changes (Modic I and II) and infection.

METHODS

Study design:

An open prospective cohort study will be performed at a single center, (Hospital Israelita Albert Einstein - HIAE) taking 1 year for recruiting, and ending 1 year after inclusion of last patient. Patients' data will be collected with a specific form created for this study. Patients will be summoned for a new magnetic resonance image of the lumbar spine one year after their surgical procedure.

All included patients will go through further treatment of ten sessions of postoperative physical therapy.

Population:

Patients who have failed conservative treatment for lumbar disc herniation undergoing lumbar decompression open surgery (microdiscectomy) will be consecutively included in the study.

Patient enrollment in the study:

Patients accepting their participation will date and sign the Informed Consent Form (ICF). After ICF is properly signed, patient will undergo an interview to complete initial demographic data and pretreatment forms.

Patient recruitment will be carried out for 24 months, when 95 patients shall be included (details of estimated n reported at sample size determination).

Patient allocation:

Patients will undergo surgery according to surgeons' preference. Attending surgeons will determine chosen operative technique according to their experience and preference.

Blinding:

Patients will not have access to the results of tissue cultures for pathogens, as well as the attending physician.

The radiologist that will analyze imaging studies of performed magnetic resonance will also be blinded to patients' data or laboratory culture results. A blinded investigator will analyze pain and function scores.

Early stopping of participation in the study:

Patients will be excluded from the study when:

* Withdrawn of ICF
* Diseased
* Patient selection flaw - incompatible eligibility criteria
* Lost to follow-up
* If patient presents clinical symptoms of infection such as severe lumbar or radicular pain, fever with no other detected foci, abnormal ESR, CRP, leucogram, and, altered imaging studies that leads to interruption of blinding of the results of culture exams.

Study stages

Sample collection:

Included patients will undergo standard fashion general anesthesia and prepped with clorhexidine solution. Intravenous antibiotics prophylaxis will be administered within first hour before skin incision, according to standard protocol of HIAE Infection Control Committee published at the hospital Pharmaceutics Manual.

Preoperative blood sample will be collected for leucogram, Erythrocyte Sedimentation Rate (ESR), and C-Reactive Protein (CRP). Same laboratory will be repeated at 1, 6 and 12 months time-point.

The excised herniated disc fragment will be immediately sent to microbiology laboratory analysis in a universal sterile container (screw cap tube) in no more than 30 minutes to be processed as follows. Same process will be applied to samples of deep muscle and ligamentum flavum at the end of the surgical procedure. Three cultures of the intervertebral disc will be done, as well as three of the ligamentum flavum and three of the multifidus muscle for each patient.

Search for pathogens:

Herniated intervertebral disc will be split in three equally sized fragments of over 2x2x5 mm and squashed in a laminar flow cabinet until homogeneous material is achieved. Same process will be carried out for the ligamentum flavum and multifidus muscle samples, although split in three fragments. Tissues will be cultured in specific growth medium and incubated according to the respective culture:

Similar criteria used by the Infectious Diseases Society of America (IDSA) to detect joint replacement infection will be adopted, which is the recommendation on at least two positive tissue cultures by the same pathogen to confirm diagnosis of infection(13).

* A - Aerobic culture For aerobic cultures, samples will be cultured in 5% sheep blood agar, chocolate agar and MacConkey agar plate, and will be placed in a 35°C incubator (CO2 atmosphere) for 5 days. If a positive bacteria culture is detected in the plate, the colony will be identified by MALDI TOF (Matrix Assisted Laser Desorption Ionization-Time of Flight) Microflex LT (Bruker Daltonics/BD).
* B - Anaerobic culture For anaerobic culture, tissue will be cultured in a Thioglycolate tube and incubated in a 35°C incubator for up to 21 days. If turbidity occurs at the Thioglycolate medium, material will be cultured in anaerobic blood agar and incubation at 35°C will be done in an anaerobic atmosphere. After growing of colonies, identification will be done by MALDI TOF.
* C - Histological analysis Anatomic pathology analysis of the other fragment of the herniated disc (2x2x5 mm) will be done. Sample will be transported in a universal container with tamponaded formalin (10%), followed by dehydration in alcohol diafanized in xylol and inclusion in paraffin (60-65°C), which will be stained in hematoxylin-eosin (HE) and GRAM staining.

  * HE: Histological cuts of 4μm will be performed, followed by clearing with xylol for 10 minutes twice, embedding with alcohol under increasing concentrations and stained with hematoxylin for 5 minutes, running water for 5 minutes, eosin for 1 minute and running water for 2 minutes followed by assembly of glass microscope slide with Entellan®.
  * GRAM: Another slide will be embedded with crystal violet for 1 minute, running water for 1 minute followed by lugol for another 1 minute and additional wash with running water. Unstaining of the slide will be done with alcohol 95% for 10 seconds followed by running water and then, stain with fuchsine for 30 seconds, running water wash again, drying and slide assembly with Entellan®.
* D - Molecular analysis of pathogens Positive cultures that present aerobic or anaerobic pathogens culturing, will be isolated and stowed refrigerated in -80°C freezer for posterior molecular analysis.

Molecular typing will be performed through Pulsed Field Gel Electrophoresis technique of isolated samples according to the protocol described by Oprica et al.(14) using Spe-I restriction enzyme and Bionumerics software for analysis of results.

Questionnaires See outcome measures

Imaging studies Magnetic resonance imaging studies will be performed in Siemens or General Electric 1.5T devices.

Lumbar disc herniation will be diagnosed through MRI in eligible patients. Included patients will be submitted to new MRI 12 months after surgery.

Two radiologists with expertise in musculoskeletal MRI will independently classify and perform measurements.

Confounding variables Data on the following confounding variables will be collected: age, gender, alcohol intake, smoking, body mass index (BMI), spinal injections with corticoid within 6 months before surgery, usage of oral corticoids up to 3 months before surgery, diabetes.

Since this information may change over time, data will be considered at time of last assessment before surgery.

Statistical planning Rate of subclinical infection (or Modic change) will be obtained by the ratio between number of positive cultures from surgical samples and total number of patients, and estimates will follow 95% confidence intervals. After infection cases are identified, we will investigate if there is an association between detected infection and patient outcomes by logistic regression models for Modic changes, ordinal logistic regression for Modic volume and size, and linear regression or general linear models for numeric outcomes, such as: low back pain, quality of life and function. All models will consider confounding variables such as: smoking and alcohol intake, diabetes, corticosteroids injection, BMI, gender, and age. Results will be presented as effects estimates such as odds ratio or mean ratio, 95% confidence intervals and p values. Study dropout cases, for any reason, will be considered for final analysis.

Sample size calculation Sample size was calculated to estimate of incidence of subclinical infection in patients with lumbar disc herniation. Considering that the rate of infection lies around 46%(3), we need to observe a minimum of 95 patients to achieve a 95% confidence interval with 10% absolute accuracy.

The necessary sample size to analyze secondary endpoints will depend on the observed rate of cases with subclinical infection in our study sample. If the observed rate is too small, an increase in the number of included patients will be needed. To better evaluate this, the sample size calculation will be revisited by the time we have reached half of initially planned sample size (48 patients).

ELIGIBILITY:
Inclusion Criteria:

* Subjects between 18 and 65 years of age; both genders; with diagnose of lumbar disc herniation undergoing open decompression surgery (microdiscectomy). Patients willing and able to go through all phases of clinical investigation and rehabilitation will be included. An Informed Consent Form (ICF) must be signed.

Exclusion Criteria:

* Patients with previous lumbar disc surgery at the same level at any point of life; patients undergoing chemotherapy; patients with any immune deficiency; patients previously submitted to disc injection and/or discography; patients submitted to previous endoscopic disc surgery; patients with fusion performed at the same stage of decompression surgery; patients with any other infection within the last six months or usage of antibiotics within the last two months; patients with incomplete specific form or data; decline to participate or sign the ICF.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with lumbar disc herniation who failed conservative treatment undergoing surgical treatment open decompression surgery (discectomy).
Sampling Method: Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2017-05-31 (Actual); Primary Completion 2019-08-15 (Actual); Study Completion 2021-05-22 (Actual)

PRIMARY OUTCOMES:
Rate of Intervertebral Disc Infection | through study completion, an average of 1 year
  The main objective of this study considers that the intervertebral disc is infected by any type of low virulence pathogen, which leads to Modic changes and chronic low back pain. Thus, calculation of the incidence of infection in lumbar disc herniations will be performed.
  1. Incidence of infection rate (IIR) will be calculated as follows: IIR = (number of detected infections) (total number of included patients)

SECONDARY OUTCOMES:
Low Back Pain | At time of patient recruitment and 1, 3, 6 and 12 months after surgical procedure
  Intensity of low back pain and limitation for daily activities of patients with and without infection will be analyzed through the Numeric Rating Score (NRS) system applied at time of patient recruitment and 1, 3, 6 and 12 months after surgical procedure. Minimal clinically important difference will be considered as an increase of 30% of baseline lumbar pain at first postoperative month, due to possible bias of postoperative pain due to surgical manipulation as well as pain due to the disc herniation itself.
EuroQoL-5D - | At timing of patient recruitment, and 1, 3, 6 and 12 months after surgery.
  Quality of life at the end of one year for both infected and uninfected groups, with and without Modic changes, will be analyzed through the validated Portuguese version of the EuroQol (EQ-5D) questionnaire. This measurement tool will be applied at timing of patient recruitment, and 1, 3, 6 and 12 months after surgery.
Function | At time of recruitment and 1, 3, 6 and 12 months after surgery.
  Function will be quantified through the Portuguese version of the Oswestry Disability Index (ODI) for lumbar pain that will be applied at time of recruitment and 1, 3, 6 and 12 months after surgery.
Modic incidence | 1 year after surgery
  Insurgent Modic changes in patients will be analyzed one year after surgery, as well as its relationship with presence or absence of infection.
  Incidence of Modic (IM) changes will be calculated for the infection group (IM infec) and for the total group (IM total) as follows:
  (number of Modic changes in infected IM infec = patients after 1 year) (total number of infections)
  IM total = number of Modic changes at final 1 year follow-up total number of patients
Volume of Modic changes | Preop and 12-month postop acquired MRI studies will be compared.
  Modic volume will be measured according to Wang et al(18). Three sagittal slices of the lumbar spine will be considered: midsagittal slice; left pedicle parasagittal slice; and right pedicle parasagittal slice. The parameters examined to quantify Modic changes will include measures of ratios of the region affected by Modic changes to the entire corresponding vertebral body, including maximal width ratio, maximal height ratio, and area ratio. Vertebral body changes will be classified accordingly to Modic changes type I, II, and III(1,2).
Adverse effects | Through study completion, an average of 1 year after inclusion
  Fail of surgical treatment (recurrence, instability, need for reoperation, etc.); need for additional physical therapy sessions; superficial infection; drainage; deep venous thrombosis; and, any other possible adverse event that may show up will be included as well.
Imaging analysis of edema | Preop and 12-month postop acquired MRI studies will be compared.
  Data will be collected for presence of vertebral or disc edema, and presence of disc hydration or not.
Imaging analysis of disc degeneration | Preop and 12-month postop acquired MRI studies will be compared.
  Disc degeneration will be collected as: normal; degeneration with height preservation; and, degeneration with loss of height. Presence of disc hydration or not.

CONTACTS AND LOCATIONS:
Overall Officials: Delio E Martins Filho, PhD, Principal Investigator — Hospital Israelita Albert Einstein
Locations (1):
- Hospital Israelita Albert Einstein, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Modic MT, Steinberg PM, Ross JS, Masaryk TJ, Carter JR. Degenerative disk disease: assessment of changes in vertebral body marrow with MR imaging. Radiology. 1988 Jan;166(1 Pt 1):193-9. doi: 10.1148/radiology.166.1.3336678.
- [Background] Modic MT, Masaryk TJ, Ross JS, Carter JR. Imaging of degenerative disk disease. Radiology. 1988 Jul;168(1):177-86. doi: 10.1148/radiology.168.1.3289089. No abstract available.
- [Background] Jensen TS, Karppinen J, Sorensen JS, Niinimaki J, Leboeuf-Yde C. Vertebral endplate signal changes (Modic change): a systematic literature review of prevalence and association with non-specific low back pain. Eur Spine J. 2008 Nov;17(11):1407-22. doi: 10.1007/s00586-008-0770-2. Epub 2008 Sep 12. PMID 18787845
- [Background] Toyone T, Takahashi K, Kitahara H, Yamagata M, Murakami M, Moriya H. Vertebral bone-marrow changes in degenerative lumbar disc disease. An MRI study of 74 patients with low back pain. J Bone Joint Surg Br. 1994 Sep;76(5):757-64. PMID 8083266
- [Background] Albert HB, Kjaer P, Jensen TS, Sorensen JS, Bendix T, Manniche C. Modic changes, possible causes and relation to low back pain. Med Hypotheses. 2008;70(2):361-8. doi: 10.1016/j.mehy.2007.05.014. Epub 2007 Jul 10. PMID 17624684
- [Background] Ohtori S, Koshi T, Yamashita M, Yamauchi K, Inoue G, Suzuki M, Takaso M, Orita S, Eguchi Y, Ochiai N, Kishida S, Kuniyoshi K, Nakamura J, Aoki Y, Ishikawa T, Arai G, Miyagi M, Kamoda H, Takahashi K. Existence of pyogenic spondylitis in Modic type 1 change without other signs of infection: 2-year follow-up. Eur Spine J. 2010 Jul;19(7):1200-5. doi: 10.1007/s00586-010-1358-1. Epub 2010 Mar 8. PMID 20213295
- [Background] Albert HB, Sorensen JS, Christensen BS, Manniche C. Antibiotic treatment in patients with chronic low back pain and vertebral bone edema (Modic type 1 changes): a double-blind randomized clinical controlled trial of efficacy. Eur Spine J. 2013 Apr;22(4):697-707. doi: 10.1007/s00586-013-2675-y. Epub 2013 Feb 13. PMID 23404353
- [Background] Albert HB, Lambert P, Rollason J, Sorensen JS, Worthington T, Pedersen MB, Norgaard HS, Vernallis A, Busch F, Manniche C, Elliott T. Does nuclear tissue infected with bacteria following disc herniations lead to Modic changes in the adjacent vertebrae? Eur Spine J. 2013 Apr;22(4):690-6. doi: 10.1007/s00586-013-2674-z. Epub 2013 Feb 10. PMID 23397187
- [Background] Stirling A, Worthington T, Rafiq M, Lambert PA, Elliott TS. Association between sciatica and Propionibacterium acnes. Lancet. 2001 Jun 23;357(9273):2024-5. doi: 10.1016/S0140-6736(00)05109-6. No abstract available. PMID 11438138
- [Background] Agarwal V, Golish SR, Alamin TF. Bacteriologic culture of excised intervertebral disc from immunocompetent patients undergoing single level primary lumbar microdiscectomy. J Spinal Disord Tech. 2011 Aug;24(6):397-400. doi: 10.1097/BSD.0b013e3182019f3a. PMID 21150662
- [Background] Carricajo A, Nuti C, Aubert E, Hatem O, Fonsale N, Mallaval FO, Vautrin AC, Brunon J, Aubert G. Propionibacterium acnes contamination in lumbar disc surgery. J Hosp Infect. 2007 Jul;66(3):275-7. doi: 10.1016/j.jhin.2007.04.007. Epub 2007 Jun 18. PMID 17573158
- [Background] Breivik H, Borchgrevink PC, Allen SM, Rosseland LA, Romundstad L, Hals EK, Kvarstein G, Stubhaug A. Assessment of pain. Br J Anaesth. 2008 Jul;101(1):17-24. doi: 10.1093/bja/aen103. Epub 2008 May 16. PMID 18487245
- [Background] Oprica C, Emtestam L, Lapins J, Borglund E, Nyberg F, Stenlund K, Lundeberg L, Sillerstrom E, Nord CE. Antibiotic-resistant Propionibacterium acnes on the skin of patients with moderate to severe acne in Stockholm. Anaerobe. 2004 Jun;10(3):155-64. doi: 10.1016/j.anaerobe.2004.02.002. PMID 16701513
- [Background] Alcohol drinking. IARC Monogr Eval Carcinog Risks Hum. 1988;44:1-378. No abstract available. PMID 3236394